CLINICAL TRIAL: NCT04271501
Title: A Prospective Blinded Randomized Within-Subject Controlled Clinical Feasibility Study to Evaluate RECELL and Melanocyte Keratinocyte Transplantation Procedure (MKTP) for Repigmentation of Stable Vitiligo Lesions
Brief Title: Feasibility Study to Evaluate RECELL and Melanocyte Keratinocyte Transplantation Procedure for Repigmentation of Stable Vitiligo Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended and Terminated to focus on CTP009 (NCT04547998) Clinical Study to Investigate the Safety and Effectiveness of RECELL for Repigmentation of Stable Vitiligo Lesions
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Device Feasibility
Other Study IDs: CTP008
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Vitiligo
Keywords: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: Each subject serves as their own control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Repigmentation will be evaluated via measurement of the area repigmented and will be rated by the patient and a Blinded Evaluator (blinded to treatment allocation) using standardized photographs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Control (No Intervention): Area without surgical intervention. Ultraviolet Lamp (UVB)
- Melanocyte-Keratinocyte Transplantation (Active Comparator): Autologous skin cell suspension prepared by laboratory based melanocyte-keratinocyte transplantation procedure technique applied to a surgically prepared area of depigmentation
  Interventions: Procedure: Melanocyte-Keratinocyte Transplantation and Ultraviolet Lamp (UVB)
- RECELL 1:5 (Experimental): Regenerative epidermal suspension diluted 1:5 applied to a surgically prepared area of depigmentation
  Interventions: Device: RECELL 1:5 and Ultraviolet Lamp (UVB)
- RECELL 1:10 (Experimental): Regenerative epidermal suspension diluted 1:10 applied to a surgically prepared area of depigmentation
  Interventions: Device: RECELL 1:10 and Ultraviolet Lamp (UVB)
- RECELL 1:20 (Experimental): Regenerative epidermal suspension diluted 1:20 applied to a surgically prepared area of depigmentation
  Interventions: Device: RECELL 1:20 and Ultraviolet Lamp (UVB)

INTERVENTIONS:
Procedure: Melanocyte-Keratinocyte Transplantation and Ultraviolet Lamp (UVB) — Application of melanocytes (aka melanocyte-keratinocyte transplantation procedure or MKTP) to surgically prepared depigmented areas
  Arms: Melanocyte-Keratinocyte Transplantation
Device: RECELL 1:5 and Ultraviolet Lamp (UVB) — Skin cell suspension dilution prepared using the RECELL System applied to a surgically prepared area of depigmentation
  Arms: RECELL 1:5
Device: RECELL 1:10 and Ultraviolet Lamp (UVB) — Skin cell suspension dilution prepared using the RECELL System applied to a surgically prepared area of depigmentation
  Arms: RECELL 1:10
Device: RECELL 1:20 and Ultraviolet Lamp (UVB) — Skin cell suspension dilution prepared using the RECELL System applied to a surgically prepared area of depigmentation
  Arms: RECELL 1:20

SUMMARY:
Prospective randomized within-subject controlled feasibility study to evaluate the clinical performance of RECELL for repigmentation of stable, depigmented lesions. The trial will evaluate 50 matched, stable depigmented areas from 10 subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible:

1. Focal, segmental or generalized (i.e., nonsegmental) vitiligo documented as stable (no new lesions nor lesions expanding in size within the preceding 12 months, regardless of whether the lesions are intended for treatment in this study).
2. The patient has not undergone topical treatment (e.g., steroids) for the study lesion within the past 60 days.
3. The patient has not undergone phototherapy (e.g., NB-UVB) for the study lesion within the past 6 months.
4. The patient is a candidate for surgical intervention for treatment of a depigmented area, defined as: the patient has been compliant but has not satisfactorily responded to topical therapy and a minimum of 3 months of phototherapy.
5. Five discrete 3cm by 3cm areas are available for treatment within the depigmented lesion.
6. The 5 study areas must be similarly sun exposed.
7. The extent of leukotrichia must be similar between the five study areas.
8. The patient is ≥ 22 years of age.
9. The patient is willing and able to comply with post-treatment at-home phototherapy and all follow-up evaluations required by the study protocol.
10. The patient agrees to abstain from any other treatment of the study areas for the duration of the his/her participation in the study (24 weeks).
11. The patient agrees to abstain from enrollment in any other interventional clinical trial for the duration of his/her participation in the study (24 weeks).
12. In the opinion of the investigator, the patient and/or guardian must be able to:

    1. Understand the full nature and purpose of the study, including possible risks and adverse events,
    2. Understand instructions, and
    3. Provide voluntary written informed consent.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible:

1. The area requiring treatment is not associated with vitiligo.
2. Study areas contain the distal phalanges.
3. The patient in unable to undergo the treatment area preparation.
4. Patients who are pregnant.
5. Patients with universalis vitiligo, depigmented areas over >30% of their body surface area, or depigmented lips and fingertips (lip-tip vitiligo).
6. Patient with a history of keloid formation.
7. Patients who have used a tanning salon in the past 60 days.
8. The patient has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives.
9. Current use of medications (e.g., anticoagulants such as such as heparin or warfarin) that in the investigator's opinion may compromise patient safety or trial objectives.
10. The patient has a known hypersensitivity to trypsin or compound sodium lactate for irrigation (Hartmann's) solution.
11. The patient has recent history (within 12 months) of Koebner phenomenon and/or confetti-like or trichrome lesions.
12. Life expectancy is less than 1 year

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Repigmentation | 24 weeks
  Percent area repigmented for each study area compared to standardized reference photos by a Blinded Evaluator

SECONDARY OUTCOMES:
Categorization of Repigmentation | 4, 12 and 24 weeks
  Categorization of each study area in terms of ranges of percent repigmentation by a Blinded Evaluator (0-25%, 26-50%, 51-79%, 80-100%)
Responders | 24 weeks
  Proportion of treated lesions achieving ≥80% or <80% repigmentation as assessed by a Blinded Evaluator.
Subject Repigmentation Rating | 4, 12 and 24 weeks
  Ratings of poor, moderate, good, or excellent
Blinded Evaluator Color Matching | 4, 12 and 24 weeks
  Assessment of color matching (0-3: poor, moderate, good, excellent) inclusive of hypopigmentation and hyperpigmentation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided